CLINICAL TRIAL: NCT07289022
Title: Evaluation of the Color Matching Ability and Clinical Success of Flowable Monochromatic and Polychromatic Composite Resins in Posterior Restorations
Brief Title: Clinical Evaluation of Flowable Monochromatic and Polychromatic Composite Resins in Posterior Restorations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Safa Tuncer, Prof. Dr., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-038
Record Dates: First submitted 2025-12-01; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dental Caries
Keywords: dental composite resin; dental caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: split-mouth
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three posterior caries lesions will be separated into three monochromatic dental composite groups (Other): Treatment of posterior caries lesions. Three of the carious lesions in the posterior four caries teeth will be separated into three groups according to material strategies described below: 1-monochromatic bulk without pigment flowable composite Omnichroma Flow Bulk (tokuyama dental) , 2-monochromatic bulk flowable composite Charisma Bulk Flow One (Kulzer), 3- monochromatic flowable composite Clearfil Majesty™ ES flow-low (Kuraray),
  Interventions: Device: dental composite
- One posterior caries lesion will be separated into one polychromatic dental flowable composite (Other): Treatment of posterior caries lesion. One of the carious lesions in the posterior four caries teeth will be separated according to the material strategies used for Grandio SO flowable polychromatic dental composite (Voco) as a control group
  Interventions: Device: dental composite

INTERVENTIONS:
Device: dental composite — Overview: Four composite resin systems will be evaluated in posterior Class II restorations for color matching ability and clinical performance over 5 years. A polychromatic composite serves as the control; three single-shade/flowable or bulk-fill composites constitute the intervention arms.
  Isolation and preparation: All restorations will be performed under rubber dam using standardized cavity preparation and finishing/polishing protocols.
  Adhesive and etching: A single adhesive approach will be used across arms per manufacturer's instructions (self etch).
  Placement:
  Control (polychromatic): Layered placement per manufacturer. Single-shade/flowable/bulk-fill arms: Incremental or bulk placement within 2-5 mm as recommended.
  Light curing: Light-emitting diode (LED) light-curing units at 1200 mW/cm² for 20 s per increment; distance and angulation standardized.
  Assessment and follow-up: Baseline, 6 months, and annually up to 5 years. Color measured with Vita Easyshade

SUMMARY:
This clinical study aims to investigate whether a single flowable composite resin system can achieve adequate color matching in posterior restorations and to compare it with a polychromatic composite system, which will serve as a control group. Clinical success will also be assessed using data obtained from the initial, six month, one-year, two-year, three-year, four-year, and five-year recall checks of the four different composite resin systems used in the study over a five-year period. L, a, and b parameters will be determined using the Vita Easyshade Compact (VITA Zahnfabrik, Bad Sackingen, Germany) Spectrophotometer device used in the study at the initial, half-year, one-year, two-year, three-year, four-year, and five-year intervals. Based on the obtained data, intraoral color changes will be determined using the CIEDE2000 color system. Each patient will be scanned with an intraoral scanner at each session. The hypothesis tested was that color matching and long-term clinical follow-up would be successful for all composite materials used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 18 years of age and have no systemic disease.
* Participants must have acceptable oral hygiene and at least 20 teeth in occlusion.
* Participants must have at least four Class I-II carious lesions requiring treatment.
* Lesions must involve both enamel and dentin, and the involved teeth must be vital and non-mobile.
* All participants must read and sign an informed consent form prior to enrollment.

Exclusion Criteria:

* Presence of any general health problem (systemic disease).
* Periodontal disease or poor oral hygiene.
* Tooth mobility or non-vital teeth in the target teeth.
* Bruxism or uncontrolled parafunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-05-05 (Estimated); Study Completion 2031-04-05 (Estimated)

PRIMARY OUTCOMES:
Clinical acceptability of restorations according to FDI criteria | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Restorations will be evaluated by a blinded assessor using the World Dental Federation (FDI) criteria across functional, esthetic, and biological domains. Clinical acceptability is defined as FDI scores 1-3. The primary analysis will report the proportion of clinically acceptable restorations and the trajectory of scores over time.

SECONDARY OUTCOMES:
Color difference (ΔE00) using the CIEDE2000 system | 1 month, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  objective color measurements will be obtained with a spectrophotometer (Vita Easyshade Compact, VITA Zahnfabrik, Bad Säckingen, Germany). L*, a*, b* values will be recorded on the restoration and adjacent tooth surfaces at each follow-up. Color difference will be calculated using the CIEDE2000 formula (ΔE00). Clinical acceptability will be defined by a predefined threshold (e.g., ΔE00 ≤ 1.8), and both mean ΔE00 and the proportion of clinically acceptable cases will be reported.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to patient confidentiality and institutional/data protection policies; aggregated results will be available in publications.

REFERENCES:
- [Background] Weick A. Issues in overturning a medical model of social work practice. Soc Work. 1983 Nov-Dec;28(6):467-71. doi: 10.1093/sw/28.6.467. No abstract available. PMID 10264483